CLINICAL TRIAL: NCT06408220
Title: OUR Stomach Health Project: A Pilot Study to Evaluate the Feasibility of Stomach Cancer Risk Assessment for Early Detection and Secondary Prevention
Brief Title: Risk Assessment Evaluation for Identifying Participants at High Risk for Stomach Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 23379; NCI-2024-03206 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23379 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-05-01; First posted 2024-05-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Biopsy; Specimen Handling; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part I (initial risk assessment) (Experimental): Participants complete questionnaires, undergo collection of a blood sample, and undergo an H. pylori breath test for gastric cancer risk assessment at baseline.
  Interventions: Procedure: Biospecimen Collection; Procedure: Breath Test; Other: Questionnaire Administration
- Part II, Cohort I (EGD, biopsy) (Experimental): Participants may undergo EGD with possible tissue biopsy within 3 months of baseline risk assessment and complete questionnaires annually up to 3 years.
  Interventions: Procedure: Biopsy; Procedure: Esophagogastroduodenoscopy; Other: Questionnaire Administration
- Part II, Cohort II (questionnaires) (Active Comparator): Participants complete questionnaires for re-assessment annually up to 3 years and may undergo EGD at year 2.
  Interventions: Procedure: Esophagogastroduodenoscopy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
  Arms: Part II, Cohort I (EGD, biopsy)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Part I (initial risk assessment)
Procedure: Breath Test — Undergo H. pylori breath test
  Arms: Part I (initial risk assessment)
Procedure: Esophagogastroduodenoscopy — Undergo EGD
  Other Names: EGD
  Arms: Part II, Cohort I (EGD, biopsy); Part II, Cohort II (questionnaires)
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial evaluates the usefulness of various risk assessment tests, including Helicobacter pylori (H. pylori) breath testing, questionnaires, and endoscopies for identifying participants at high risk for stomach cancer. H. pylori is a bacteria that causes stomach inflammation and ulcers in the stomach. People with H. pylori infections may be more likely to develop cancer in the stomach. H. pylori breath testing can help identify the presence of H. pylori infection in a participant and help identify if the participant may be at a higher risk of developing stomach cancer. An endoscopy uses a thin, flexible lighted tube that is inserted inside the esophagus, stomach, and first part of the small intestine. This allows the doctor to see and look for abnormal areas that may need to be biopsied. Risk assessment including H. pylori evaluation, questionnaires, and endoscopies may help identify participants at high risk for stomach cancer and may be a useful screening tool for earlier stomach cancer diagnosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of using community outreach and clinical assessment to identify persons at high risk for gastric cancer.

SECONDARY OBJECTIVES:

I. To determine the presence of gastric cancer (GC) associated risk factors amongst the diverse ethnic populations (in greater Orange and Los Angeles Counties).

II. To determine the proportion of high-risk patients who are willing to undergo upper endoscopy.

III. To identify actionable diagnoses on upper endoscopy of high-risk individuals.

EXPLORATORY OBJECTIVE:

I. To assess population-based understanding of gastric cancer.

OUTLINE:

PART I: Participants complete questionnaires, undergo collection of a blood sample, and undergo an H. pylori breath test for gastric cancer risk assessment at baseline.

PART II: High-risk participants are assigned to cohort I and non-high risk participants are assigned to cohort II.

COHORT I: Participants may undergo esophagogastroduodenoscopy (EGD) with possible tissue biopsy within 3 months of baseline risk assessment and complete questionnaires annually up to 3 years.

COHORT II: Participants complete questionnaires for re-assessment annually up to 3 years and may undergo EGD at year 2.

Participants are followed up annually for a total of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 40 years to ≤ 80 years
* Identify as a racial minority either Asian, Hispanic, or Black American
* Willingness to:

  * Provide blood samples and undergo upper endoscopy

Exclusion Criteria:

* Identify as Non-Hispanic White
* History of gastric cancer
* Known premalignant lesions of the stomach
* History of upper endoscopy within 2 years
* Women of childbearing potential: Pregnant/ nursing
* An employee who is under the direct/indirect supervision of the principal investigator (PI)/a coinvestigator/the study manager
* A direct study team member

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of screening individuals found to be at high risk for gastric cancer (feasibility) | At time of screening up to 3 years
  Study feasibility will be defined as ≥ 10% of screened individuals found to be at high risk for gastric cancer. The study will be successful if ≥ 10% of screened individuals (24 of ≤ 240) have a risk score of ≥ 12 or have signs/symptoms that have persisted for ≥ 1 month that are associated with gastric cancer. The reported results will include counts/proportions of screened individuals found to be at high risk for gastric cancer (≥ 12 risk score).

CONTACTS AND LOCATIONS:
Overall Officials: Yanghee Woo, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States